CLINICAL TRIAL: NCT05518474
Title: Effectiveness of Self-proning and Repositioning in Outpatients With COVID-19: a Randomized Controlled Internal Pilot Trial
Brief Title: Self-proning and Repositioning in COVID-19 Outpatients at Risk of Complicated Illness
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient participant enrollment due to dwindling case numbers/case severity
Sponsor: Unity Health Toronto (Other)
Collaborators: Applied Health Research Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: homeproningpilot_21_069
Record Dates: First submitted 2022-08-22; First posted 2022-08-26 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: COVID-19; COVID-19 Pneumonia; Proning; Hospitalization; Death; Outpatient; Complication
MeSH Terms: conditions — COVID-19; Death

STUDY DESIGN:
Intervention Model Description: Open label, pragmatic, randomized controlled internal pilot trial (vanguard phase)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-proning (Experimental): Participants assigned to the intervention arm will receive a SMS link to a PDF containing instructions on proning/repositioning and information about its physiological benefits. They'll also receive a PDF with standard recommendations for treating COVID-19 at home. Participants will be encouraged to lie flat on their belly, on their side, or sit upright and rotate between these positions when lying down during the day and night. Participants will be sent a daily SMS "proning reminder" and asked to complete a secure REDCap survey regarding their proning activity. They'll be advised to prone and reposition for seven days minimum whenever they are lying down. Participants who have failed to reach their functional baseline after this time period will be advised to continue doing so. Follow up assessment by telephone will be conducted in 7 day increments from baseline up to 28 days.
  Interventions: Other: Self-proning
- Standard care (No Intervention): Participants assigned to the comparator arm will receive a SMS link to a PDF with standard recommendations for treating COVID-19 at home. This includes antipyretics and analgesics for fever, myalgias, and headaches; hydration; and rest with advancement of activity as soon as tolerated. Follow up assessment by telephone will be conducted in 7 day increments from baseline up to 28 days.

INTERVENTIONS:
Other: Self-proning — Rotating between lying flat with the chest down, on one's side or sitting up every 30 minutes to 2 hours when lying down during the day or while sleeping at night.
  Other Names: Self-proning/repositioning; Home-proning
  Arms: Self-proning

SUMMARY:
The rapid development of safe and effective COVID-19 treatment is a global health priority. Numerous studies evaluating therapies for this disease are currently underway, but the majority of these are in hospitalized patients with severe illness. Consequently, there is an urgent need to identify therapies that prevent mild COVID-19 cases in the community from becoming more severe. "Proning" or lying face down in bed has been shown to improve breathing and oxygen levels in COVID-19 patients, reducing the need for breathing tubes and ventilators and increasing survival. The current study will investigate whether proning and repositioning (lying on one's side or sitting up) can prevent mild cases of COVID-19 from becoming more severe resulting in fewer hospitalizations and death. A randomized controlled trial will be used to reduce the risk of bias when testing this intervention. Unvaccinated or partially vaccinated adult patients with a positive COVID-19 test willing to participate and well enough to be treated outside the hospital will be randomly assigned to one of two groups: a home-proning intervention group with instructions and daily reminders to prone and reposition during the day and at night, and a standard care group. Our goal is to assess whether home-proning/repositioning leads to fewer hospitalizations and death when compared with standard care. We'll also compare recovery time, use of antibiotics and follow up emergency department visits between these two groups. The current pilot study will assess the feasibility of a larger investigation or "main trial", meaning it will be small scale test of methods and procedures to be used on a larger scale.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Positive SARS-CoV-2 PCR test
3. Presence of two or more of the following criteria:

   1. Age>55 years
   2. Fever by history or at presentation
   3. Cough
   4. Dyspnea/shortness of breath
   5. Fatigue necessitating daytime bed rest
   6. One or more of the following medical conditions:

      * Hypertension
      * Diabetes
      * Cardiovascular disease
      * Chronic lung disease
      * Chronic kidney disease
      * Obesity (BMI≥30kg/m2)
   7. Tachycardia > 110 bpm
   8. Oxygen saturation <94%
   9. One or more of the following laboratory abnormalities:

      * Lymphocytes <1500/microL
      * ESR > 100 mm/h
      * CRP > 10 mg/L
      * D-Dimer > 1000 ng/mL
      * LDH > 240 U/L
   10. Bilateral infiltrates or ground glass opacities on chest x-ray or CT scan
4. Socially and medically fit for discharge
5. Access to a smartphone

Exclusion Criteria:

1. Pregnancy >20/40 weeks
2. Body mass index (BMI) >40 kg/m2.
3. Skeletal deformities that interfere with proning
4. Developmental delay or cognitive impairment that would preclude patient cooperation
5. Other contraindications to proning including any of the following: recent abdominal surgery, active vomiting, acute intoxication.
6. Unlikely to adhere to the proning protocol according to the treating physician's judgment
7. Fully vaccinated for COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Composite of hospitalization and all cause mortality | Up to 28 days post-randomization
  The primary outcome is a composite of hospital admission and all-cause mortality. This will be ascertained using telephone follow up and deterministic record linkage performed by the Institute for Clinical Evaluative Sciences (ICES) using their Discharge Abstract Database (DAD).

SECONDARY OUTCOMES:
Hospitalization | Up to 28 days post-randomization
All cause mortality | Up to 28 days post-randomization
Time to functional recovery in days | Up to 28 days post-randomization
  Defined as: resolution of fever for 48 hours, significant symptom reduction and ability to perform most daily activities or return to work, if applicable, for two consecutive days.
Use of antibiotics for respiratory illness | Up to 28 days post-randomization
Follow up emergency department assessment without hospital admission | Up to 28 days post-randomization
  Number of subsequent emergency department visits by study participants that relate to the initial COVID-19 presentation but do not result in hospital admission

OTHER OUTCOMES:
Feasibility outcome: successful recruitment | Through study completion, on average one year
  Defined as >=50% of eligible participants agreeing to enrollment
Feasibility outcome: successful retention of trial participants, | Up to 28 days
  Defined as <10% attrition rate
Feasibility outcome: adherence to the intervention | Up to 28 days
  Defined as self-proning and repositioning daily for >=75% of days of symptom duration. Adherence will be ascertained through daily survey of study participants.

CONTACTS AND LOCATIONS:
Locations (1):
- St. Joseph's Health Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF